CLINICAL TRIAL: NCT02982447
Title: Comparison of Detection and Miss Rates of Colorectal Adenoma by Blue Laser Imaging (BLI) Versus Conventional White Light Colonoscopy.
Brief Title: Comparison of Detection and Miss Rates of Blue Laser Imaging Versus Conventional White Light Colonoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yangzhou No.1 People's Hospital (Other)
Responsible Party: Principal Investigator, zhi jie-hua, Principal Investigator, Yangzhou No.1 People's Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Yangzhou1PH
Record Dates: First submitted 2016-11-19; First posted 2016-12-05 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Colorectal Adenoma
Keywords: blue laser imaging,detection,randomized trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Blue Laser Imaging colonoscopy (Active Comparator): Insertion to cecum was performed under white light(WL) and once the cecum was reached, the Blue Laser Imaging mode was switched on during withdrawal of endoscope for complete colonic examination. Second colonoscopic examination was performed in a similar manner after the first complete withdrawal of the colonoscope. WL was used on insertion and WL was used on withdrawal
  Interventions: Device: blue laser imaging colonoscopy
- conventional white light colonoscopy (Experimental): In this arm, WL was used for both insertion and withdrawal of the colonoscope during the first-pass and second-pass examinations.
  Interventions: Device: conventional white light colonoscopy

INTERVENTIONS:
Device: blue laser imaging colonoscopy — Insertion to cecum was performed under white light(WL) and once the cecum was reached, the Blue Laser Imaging mode was switched on during withdrawal of endoscope for complete colonic examination. Second colonoscopic examination was performed in a similar manner after the first complete withdrawal of the colonoscope. WL was used on insertion and WL was used on withdrawal
  Arms: Blue Laser Imaging colonoscopy
Device: conventional white light colonoscopy — In this arm, WL was used for both insertion and withdrawal of the colonoscope during the first-pass and second-pass examinations.
  Arms: conventional white light colonoscopy

SUMMARY:
It is a randomized controlled trial with tandem colonoscopy.Participants were randomized for use of either blue laser imaging or conventional White Light Colonoscopy on withdrawal method.comparison of detection and miss rates of BLI group Versus conventional White Light Colonoscopy.

DETAILED DESCRIPTION:
blue laser imaging (BLI) are a new imaging systems used in endoscopy which are recently developed. According to three recently published reports, the diagnostic ability of adenoma characterization using blue laser imaging compares favorably with narrow band imaging. No published data are available to date regarding adenoma detection with blue laser imaging.BLI has the possibility to increase the detection of colorectal polyps by sufficient brightness and clearer endoscopic images.The investigators recruited participants who underwent colonoscopy for symptoms,screening,or surveillance.Participants were randomized for use of either blue laser imaging (BLI) or conventional white light colonoscopy on withdrawal method.Lesions detected on first-pass and second-pass examination were used for adenoma detection and miss rates,respectively.The primary outcomes is to compare the adenoma and poly detection rates of BLI with conventional white light Colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* consecutive patients who were underwent colonoscopy in our center for diagnostic work up of colonic symptoms,surveillance of colorectal polyps, and colorectal cancer screening.

Exclusion Criteria:

* history of colon cancer, colectomy familial adenomatous polyposis, or inflammatory bowel diseases;
* severe intestinal stenosis or obstruction;coagulation，disorders;
* pregnancy;
* and colonoscopy examinations with inadequate bowel cleanliness

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-04 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
comparison of colorectal adenoma detection rates of blue laser imaging (BLI) Versus conventional White Light Colonoscopy | 6 months
comparison of colorectal adenoma miss rates of blue laser imaging (BLI) Versus conventional White Light Colonoscopy | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: zhi jie hua, postgraduate, Principal Investigator — First People's Hospital of Yangzhou
Locations (1):
- First people's hospital of yangzhou, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yoshida N, Hisabe T, Inada Y, Kugai M, Yagi N, Hirai F, Yao K, Matsui T, Iwashita A, Kato M, Yanagisawa A, Naito Y. The ability of a novel blue laser imaging system for the diagnosis of invasion depth of colorectal neoplasms. J Gastroenterol. 2014 Jan;49(1):73-80. doi: 10.1007/s00535-013-0772-7. Epub 2013 Mar 15. PMID 23494646
- [Result] Yoshida N, Yagi N, Inada Y, Kugai M, Okayama T, Kamada K, Katada K, Uchiyama K, Ishikawa T, Handa O, Takagi T, Konishi H, Kokura S, Yanagisawa A, Naito Y. Ability of a novel blue laser imaging system for the diagnosis of colorectal polyps. Dig Endosc. 2014 Mar;26(2):250-8. doi: 10.1111/den.12127. Epub 2013 Jun 3. PMID 23731034
- [Result] Togashi K, Nemoto D, Utano K, Isohata N, Kumamoto K, Endo S, Lefor AK. Blue laser imaging endoscopy system for the early detection and characterization of colorectal lesions: a guide for the endoscopist. Therap Adv Gastroenterol. 2016 Jan;9(1):50-6. doi: 10.1177/1756283X15603614. PMID 26770267